CLINICAL TRIAL: NCT03488771
Title: Evaluation of Cell-mediated Immune Response by QuantiFERON Monitor® Assay in Kidney Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Hospital Merkur (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Sponsor
Other Study IDs: CHMerkurQFM
Record Dates: First submitted 2018-03-22; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Kidney Transplant Infection; Kidney Transplant Rejection
Keywords: kidney transplantation; rejection; infection; immunosuppression
MeSH Terms: conditions — Rejection, Psychology; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Kidney transplant recipients without clinical/laboratory/biopsy signs of infection or graft rejection
- Infection: Kidney transplant recipients presenting with clinical or laboratory signs of infection (bacterial or viral)
- Rejection: Kidney transplant recipients presenting with clinical, laboratory or biopsy signs of graft rejection.

SUMMARY:
All kidney transplant recipients require immunosuppression, the net level of which is difficult to assess. Current practice in assessing immune reactivity is to monitor levels of some immunosuppressive drugs. QuantiFERON Monitor® (QFM) is an in vitro diagnostic test that detects interferon-γ (IFN-γ) release in peripheral blood. Its clinical utility in assessment of the net state of immunosuppression in kidney transplant recipients has not been well studied. The aim of our study is to evaluate the discriminating value of QFM testing results for infection and rejection in a single-centre cohort of kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Kidney/Liver kidney/Simultaneous pancreas and kidney transplantation

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-03-05 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Infection | throughout the study period (Kidney transplant recipients from 1 day date of tx to 15 years after tx)
  Interferon gamma level in patients with infection

SECONDARY OUTCOMES:
Rejection | throughout the study period (Kidney transplant recipients from 1 day date of tx to 15 years after tx)
  Interferon gamma levels in patients with rejection

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Merkur, Zagreb, HR, Croatia